CLINICAL TRIAL: NCT04555005
Title: Implementation of a Mindfulness-based Crisis Intervention for Frontline Healthcare Workers During the COVID-19 Outbreak in a Public General Hospital in Madrid, Spain
Brief Title: Mindfulness-based Crisis Intervention for COVID-19 Frontline Healthcare Workers During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Mind-COVID-19
Record Dates: First submitted 2020-06-11; First posted 2020-09-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Mindfulness; COVID-19; Healthcare Worker
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindfulness based intervention (Other): Mindfulness based intervention for frontline healthcare workers during COVID-19 outbreak
  Interventions: Other: Mindfulness based intervention

INTERVENTIONS:
Other: Mindfulness based intervention — Mindfulness based intervention for frontline healthcare workers during COVID-19 outbreak

SUMMARY:
The COVID-19 outbreak is having an impact on the well-being of healthcare workers. Previous reports on pandemics show that such an impact may last beyond the time of the outbreak. Mindfulness-based interventions help healthcare professionals to reduce stress and may foster resilience and recovery, although they have never been tested in a context such as the current one. This single-arm trial explores the acceptability, safety and usefulness of an on-site, brief Mindfulness-based intervention to reduce stress for front line health workers during a crisis.

ELIGIBILITY:
Inclusion Criteria:

* All frontline healthcare workers present in the ward at the time of intervention

Exclusion Criteria:

* Extreme adverse events

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-04-26 (Actual)

PRIMARY OUTCOMES:
Perceived helpfulness to reduce current stress | through study completion, up to three days
  The outcome was measured by a 10-point visual analogue scale developed for this study, where 0 was "it did not help me at all" and 10 was "it helped me a lot".

CONTACTS AND LOCATIONS:
Locations (1):
- La Paz University Hospital, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez-Vega B, Palao A, Munoz-Sanjose A, Torrijos M, Aguirre P, Fernandez A, Amador B, Rocamora C, Blanco L, Marti-Esquitino J, Ortiz-Villalobos A, Alonso-Sanudo M, Cebolla S, Curto J, Villanueva R, de-la-Iglesia MJ, Carracedo D, Casado C, Vidal E, Trigo D, Iglesias N, Cabanas D, Mellado L, Garcia D, Fernandez-Encinas C, Navarro R, Mediavilla R, Vidal-Villegas MP, Bravo-Ortiz MF, Bayon C. Implementation of a Mindfulness-Based Crisis Intervention for Frontline Healthcare Workers During the COVID-19 Outbreak in a Public General Hospital in Madrid, Spain. Front Psychiatry. 2020 Oct 30;11:562578. doi: 10.3389/fpsyt.2020.562578. eCollection 2020. PMID 33329103